CLINICAL TRIAL: NCT03410329
Title: Comparison of the Effect of Different Frequencies Weekly Training on Body Composition, Cardiometabolic Risk Factors and Handgrip Strength in Overweight and Obese Women
Brief Title: Effect of Different Frequencies Weekly Training in Overweight/Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francesco Campa (Other)
Responsible Party: Sponsor-Investigator, Francesco Campa, Principal Investigator, University of Bologna
Organization: University of Bologna (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12022016
Record Dates: First submitted 2018-01-12; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Sensitivity Training Groups
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High weekly training frequency (Experimental): three sessions a week of resistance training
  Interventions: Other: Resistance training
- Low weekly training frequency (Experimental): one workouts per week
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — Physical activity

SUMMARY:
The aim of this study was to evaluate the effects of a resistance training programme of one or three times a week on body composition, cardiometabolic risk factors and handgrip strength in overweight and obese women

DETAILED DESCRIPTION:
This study aimed to determine the effects of supervised structured 6 months resistance training and a restricted caloric diet on body composition, cardiometabolic risk factors and handgrip strength in overweight and obese women. 45 women were randomly assigned to one of two groups: a group with a high-weekly frequency of three times a week (HIGH) and a group that performed only one weekly session (LOW).HbA1c, percentage of fat mass and handgrip strength were taken before and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

overweight or obese

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Fat mass | 24 weeks
  anthropometric measurements

SECONDARY OUTCOMES:
Handgrip strength | 24 weeks
  mechanical dynamometer

OTHER OUTCOMES:
HbA1c | 24 weeks
  It was measured by exchange high-performance liquid chromatograph using standardised laboratory procedures

IPD SHARING:
Plan to Share IPD: Undecided